CLINICAL TRIAL: NCT03983577
Title: Efficacy of Point Of Service Testing in Metastatic Breast Cancer
Brief Title: Efficacy of Point Of Service Testing in MBC
Acronym: EPOST MBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ePOST
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Cancer; Breast Cancer
Keywords: genetic counseling
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Point of service delivery model (Experimental): After the informed consent is signed, the participant will watch a standardized video on the principles of genetic testing. At the end of the video, the provider will return to answer any remaining questions. The participant will receive pre- and post- surveys for evaluation of the delivery model.
  Interventions: Other: Point of service delivery model

INTERVENTIONS:
Other: Point of service delivery model — Participants will receive the pre-test survey, followed by the combined provider/telehealth genetic counseling education video for genetic testing. Afterwards, the participants will receive a post-test and patient satisfaction survey.

SUMMARY:
This study will assess the efficacy of an innovative point of service cancer genetics counseling delivery model for metastatic breast cancer (MBC) patients whom have received a referral for hereditary cancer genetic counseling and testing.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent.
* Able to speak and read in the English language.
* Have a diagnosis of human epidermal growth factor receptor 2 (HER2) negative metastatic breast cancer.
* Participants must be enrolled in the parent registry study.

Exclusion Criteria:

* Genetic testing for a breast cancer gene (BRCA) BRCA1 and BRCA2 mutation completed after 2013 or any BRCA 1 and BRCA2 testing with large rearrangement testing. Prior genetic counseling is allowed.
* Psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients/participants that undergo hereditary cancer genetic testing after the telehealth intervention. | 24 months
  Defined as the number of participants who opt to undergo hereditary cancer genetic testing as a percentage of the total number of participants enrolled.

SECONDARY OUTCOMES:
Overall participant satisfaction | 24 months
  Patient satisfaction will be assessed with an adapted Genetic Counseling Satisfaction Scale (aGCSS). Each item is scored from 1- 5, with 1 being strongly disagree and 5 being agree strongly. The scores are added then divided by 5 to give a mean score.
Clinical decisional conflict score | 24 months
  Decisional conflict will be assessed using the Decisional Conflict Scale (Sure Test Version). The 4 items are summed. Scores range from 0 (extremely high decisional conflict) to 4 (no decisional conflict). A score of less than or equal to 3 indicates decisional conflict.
Overall participant anxiety | 24 months
  Participant anxiety will be assessed with the Hospital Anxiety and Depression Scale (HADS-Anxiety scale). Each item is scored between 0- 3 with a total score between 0- 21 possible. Scores of 0-7 indicates normal; scores of 8-10 indicates borderline abnormal; scores of 11-21 indicates abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Nye, MD, Principal Investigator — University of Kansas
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States